CLINICAL TRIAL: NCT02152007
Title: Phase 1b Clinical Trial Using Topical Sirolimus for the Treatment of Pachyonychia Congenita
Brief Title: Topical Sirolimus for the Treatment of Pachyonychia Congenita (PC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransDerm, Inc. (Industry)
Collaborators: Pachyonychia Congenita Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TD201 - CS01; FD-R-05116 (Other Grant/Funding Number: Orphan Products Development (OPD)); NCT02057614 (obsolete NCT alias)
Record Dates: First submitted 2014-02-05; First posted 2014-06-02 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Pachyonychia Congenita
Keywords: pachyonychia congenita
MeSH Terms: conditions — Pachyonychia Congenita

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Split-body 1% sirolimus cream (TD201 1%) (Experimental): This is a split-body design. Subjects will self-administer 1% topical sirolimus cream or placebo cream (no drug, vehicle control) on the plantar surface of each foot. At least one foot will be treated with topical sirolimus at some time during the study. Application will be one time daily for a total of 26 weeks. There will be an additional follow-up visit 3 months after the last application of study drug. The total duration of the study is 39 weeks.
  Interventions: Drug: 1% sirolimus cream (TD201 1%)

INTERVENTIONS:
Drug: 1% sirolimus cream (TD201 1%) — 1% sirolimus cream (TD201 1%)

SUMMARY:
A study to evaluate safety and efficacy of topical sirolimus to treat plantar keratoderma in adults with PC. Subjects may receive either placebo or treatment with at least 1 foot receiving topical sirolimus at some time. For certain phases of the study treatment assignment to the right and left foot will be randomized in a double blind fashion. Blood levels will test systemic absorption of sirolimus. Other safety and efficacy measures will be taken through the 39-week study duration. Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* Be capable of understanding the purpose and risks of the study and sign a written Informed Consent Form (ICF)
* Be male or female ≥ 16 years of age at the time of the screening visit
* Have a confirmed diagnosis of PC by genotyping (e.g., familial) and clinically correlated painful keratoderma.
* Have roughly symmetrical calluses of similar severity on the plantar surface of both feet
* Women of childbearing potential must have a negative serum pregnancy test
* Subjects, whether male or female, with reproductive potential and who are sexually active must agree to use double-barrier contraception methods

Exclusion Criteria:

A Subject with any of the following criteria is not eligible for inclusion in this study:

* Use of other investigational drugs within 30 days of the screening visit and/or has not recovered from any side effects of prior investigational drugs or procedure in the affected area (e.g., a biopsy)
* Significant condition in the dermatologic treatment area such as trauma, or nonhealing chronic wound
* Pregnant or nursing (lactating) female, or a positive serum pregnancy test
* Active infection either systemic or local near the site of treatment requiring chronic or prolonged use of antimicrobial agents
* Known immunodeficiency including: Hepatitis A; Hepatitis B; Hepatitis C; Human Immunodeficiency Virus (HIV)

Prior and Current Treatment

* Unable to be discontinued from drugs known to either be inducers or inhibitors of CYP3A4/5 enzymes
* Unable to be discontinued from drugs known to be P-glycoprotein inhibitors

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Kaspar, PhD, Study Chair — TransDerm, Inc.
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Split-body 1% Sirolimus Cream (TD201 1%)
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This is a split-body design. After a 2-week run in phase in which both feet were treated with placebo, feet were randomized and one foot received 1% sirolimus and the other placebo ("randomized phase") for 8 weeks. Following the randomized phase, patients applied 1% sirolimus to both feet ("open label phase") for an additional 8 weeks.
Arm/Group | Split-body 1% Sirolimus Cream (TD201 1%)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Systemic Absorption Through Measurement of Serum Sirolimus Trough Levels
Description: The primary outcome measure for this Phase 1b safety study is evaluation of system absorption through measurement of serum sirolimus trough levels. The limit of detection of the assay was 2.0 ng/mL.
Time Frame: Two weeks and every 1-2 months for 24 weeks or within 2 weeks after the last dose of study drug
Population: Starting at week 13, visit 4, there were only 14 participants with available data.
Measure: Number; unit: participants
Arm/Group | Split-body 1% Sirolimus Cream (TD201 1%)
Number analyzed (Participants) | 15
participants
  Visit 1, Baseline, <2.0 ng/mL | 15
  Visit 2, Week 3, <2 ng/mL | 15
  Visit 3, Week 7, <2 ng/mL | 15
  Visit 4, Week 13, <2 ng/mL | 14
  Visit 5, Week 17, <2 ng/mL | 14
  Visit 6, Week 25, <2 ng/mL | 14
  Visit 7, Week 37, <2 ng/mL | 14

2. Secondary Outcome: Weekly Assessments Recorded in the PC Quality of Life Index
Description: Patient-reported weekly assessment in the PC Quality of Life Index
Time Frame: Weekly for 39 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Daily Assessments Recording in the PC Measurement Diary
Time Frame: Weekly for 39 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Investigator Assessment of Local Tolerability
Description: Investigator assessment of local tolerability at the application sites on the plantar surfaces will be evaluated by the Investigator according to a 4-point scale (0, 1, 2, or 3; none to severe) with regard to: erythema, pruritis, stinging/burning, and crusting/erosion
Time Frame: Prior to application of study drug and within 15-45 minutes after application of study drug at each visit for 39 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Cream (Vehicle Control): Placebo Cream (Vehicle Control)
Arm/Group | Split-body 1% Sirolimus Cream (TD201 1%) | Placebo Cream (Vehicle Control)
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 Pre, Erythema Score (0-3) | 0.2 (0.41) | 0.2 (0.41)
  Visit 1 Pre, Pruritus Score (0-3) | 0.1 (0.26) | 0 (0)
  Visit 1 Pre, Stinging/Burning (0-3) Score | 0 (0) | 0.1 (0.26)
  Visit 1 Pre, Crusting/Erosion Score (0-3) | 0.1 (0.26) | 0.1 (0.26)
  Visit 1 Post, Erythema Score (0-3) | 0.2 (0.41) | 0.2 (0.41)
  Visit 1 Post, Pruritus Score (0-3) | 0 (0) | 0 (0)
  Visit 1 Post, Stinging/Burning Score (0-3) | 0 (0) | 0.1 (0.26)
  Visit 1 Post, Crusting/Erosion Score (0-3) | 0.1 (0.26) | 0.1 (0.26)
  Visit 4 Pre, Erythema Score (0-3) | 0 (0) | 0 (0)
  Visit 4 Pre, Pruritus Score (0-3) | 0.1 (0.28) | 0.1 (0.28)
  Visit 4 Pre, Stinging/Burning Score (0-3) | 0.1 (0.28) | 0 (0)
  Visit 4 Pre, Crusting/Erosion Score (0-3) | 0.1 (0.28) | 0.2 (0.38)
  Visit 4 Post, Erythema Score (0-3) | 0 (0) | 0 (0)
  Visit 4 Post, Pruritus Score (0-3) | 0 (0) | 0 (0)
  Visit 4 Post, Stinging/Burning Score (0-3) | 0.1 (0.28) | 0 (0)
  Visit 4 Post, Crusting/Erosion Score (0-3) | 0.1 (0.28) | 0.2 (0.38)
  Visit 7 Pre, Erythema Score (0-3) | 0.2 (0.58) | 0.2 (0.58)
  Visit 7 Pre, Pruritus Score (0-3) | 0.2 (0.58) | 0.2 (0.58)
  Visit 7 Pre, Stinging/Burning Score (0-3) | 0.3 (0.61) | 0.3 (0.61)
  Visit 7 Pre, Crusting/Erosion Score (0-3) | 0.4 (0.65) | 0.3 (0.61)

5. Other Pre Specified Outcome: Standardized Photographs
Description: An expert in the disease who is blinded to the study treatment will read the photographs of the callus area taken at each study visit. The reader will assess changes to the calluses based on criteria such as blisters, cracks, small/large size, and red or bloody spots on the callus. Change in calluses will be reported for both the right and left foot.
Time Frame: Each study visit over 39 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of the study, up to 39 weeks
Arm/Group | Split-body 1% Sirolimus Cream (TD201 1%)
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Split-body 1% Sirolimus Cream (TD201 1%) (N=15)
Nausea (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was primarily concerned with safety endpoints. Efficacy endpoints need to be improved for follow on studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No